CLINICAL TRIAL: NCT02191826
Title: Study of SOM0226 in Familial Amyloid Polyneuropathy (FAP) Patients and Asymptomatic Carriers to Evaluate Protein Stabilization Activity
Brief Title: Study of SOM0226 in Familial Amyloid Polyneuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SOM Innovation Biotech SA (Industry)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOMCT01-C; 2014-001586-27 (EudraCT Number)
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Familial Amyloid Polyneuropathy (FAP)
Keywords: Transthyretin; TTR; Amyloidosis; SOM0226; Familiar Amyloid Polyneuropathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis | interventions — Tolcapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOM0226 single dose (Experimental)
  Interventions: Drug: SOM0226
- SOM0226 multiple doses (Experimental)
  Interventions: Drug: SOM0226

INTERVENTIONS:
Drug: SOM0226 — Oral

SUMMARY:
Clinical proof of concept study to evaluate SOM0226 efficacy in TTR Amyloidosis.

DETAILED DESCRIPTION:
This is an open label interventional Phase IIa proof of concept clinical trial designed in two phases separated by a washout period of 6 weeks (± 2 weeks) , to evaluate the TTR stabilization activity of SOM0226 in healthy volunteers (wild type), TTR-FAP patients and asymptomatic carriers.

* Phase A (24 hours): SOM0226 single dose
* Phase B (32 hours): SOM0226 multiple dose

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above at the time of consent
* Two cohorts defined by TTR variant (wild type: healthy volunteers; TTR mutant: asymptomatic carriers with documented mutation in TTR or diagnosed TTR-FAP patients (stage 1 or 2) not undergoing pharmacological treatment with Vyndaqel
* Body Mass Index (BMI) > 17.5 kg/m2
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 2 month thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study
* Evidence of history of clinically significant hepatic disease
* An ALT or AST measurement > 2 times the ULN (Upper Limit of Normal)
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Donation of blood during the study or within the past 4 weeks
* Treatment (during the study or within the past 4 weeks) with a prescription or investigational drug for the treatment of TTR amyloidosis
* Treatment with NSAIDs (nonsteroidal antiinflammatory drug) during the study or within the past 4 weeks. The following NSAID are allowed: acetylsalicylic acid, etodolac, ibuprofen, indomethacin, ketoprofen, nabumetone, naproxen, nimesulide, piroxicam and sulindac

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
TTR stabilization | 24 hours and 32 hours
  TTR stabilization will be measured by determining the concentration of tetrameric TTR after denaturation. The ratio of TTR tetramer after denaturation / TTR tetramer before denaturation of plasma samples from treated subjects will be compared to their baseline ratio. TTR stabilization will be determined as percentage of the baseline ratio.

SECONDARY OUTCOMES:
Pharmacodynamics assessment | 24 hours and 32 hours
  Determine the minimal molar ratio SOM0226:TTR that must be reached in plasma to confer maximal TTR stabilization
Safety | 24 hours
  Drug safety will be assessed by blood biochemistry and hematology analysis, patient exploration and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Josep Gámez, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Gamez J, Salvado M, Reig N, Sune P, Casasnovas C, Rojas-Garcia R, Insa R. Transthyretin stabilization activity of the catechol-O-methyltransferase inhibitor tolcapone (SOM0226) in hereditary ATTR amyloidosis patients and asymptomatic carriers: proof-of-concept study. Amyloid. 2019 Jun;26(2):74-84. doi: 10.1080/13506129.2019.1597702. Epub 2019 May 23. PMID 31119947
- See also: Related Info — http://www.sombiotech.com